CLINICAL TRIAL: NCT01680575
Title: Development of a Risk Model Predicting Chemotherapy-induced Grade 3-4 Neutropenia by Paclitaxel/Carboplatin in Epithelial Ovarian Cancer: Prospective Observational Study for Model Development and Retrospective Study for Validation of Developed Model
Brief Title: Study on Neutropenia Induced by Adjuvant Paclitaxel/Carboplatin Chemotherapy in Patients With Epithelial Ovarian Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Jeong-Yeol Park, Clinical Assistant Professor, Asan Medical Center
Other Study IDs: NEPACA-OVCA
Record Dates: First submitted 2012-09-04; First posted 2012-09-07 (Estimated); Last update posted 2017-05-31 (Actual); Status verified 2017-05

CONDITIONS: Epithelial Ovarian Cancer
Keywords: Neutropenia; Paclitaxel; Carboplatin; Epithelial ovarian cancer
MeSH Terms: conditions — Carcinoma, Ovarian Epithelial; Neutropenia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Training cohort: This cohort is a prospective cohort to develop a risk prediction model. This cohort include patients who underwent staging operation or debulking operation for epithelial ovarian cancer and are planned to receive ajuvant chemotherapy with paclitaxel/carboplatin up to 6 cycles.
- Validation cohort: This is a retrospective cohort for validation of a risk prediction model developed using training cohort.
  This is consisted with 600 patients with epithelial ovarian cancer who received adjuvant chemotherapy with paclitaxel/carboplatin after staging operation or debulking operation.

SUMMARY:
To develop a robust prediction model to predict the occurrence of grade 3-4 neutropenia induced by adjuvant paclitaxel/carboplatin chemotherapy in patients with epithelial ovarian cancer and to validate this model.

ELIGIBILITY:
Inclusion Criteria:

* Patients with FIGO stage I-IV epithelial ovarian cancer after staging or debulking surgery
* Patients who is planned to receive (prospective cohort) ro who received (retrospective cohort) adjuvant chemotherapy with paclitaxel and carboplatin
* Patients who have signed approved informed consent

Exclusion Criteria:

* Uncontrolled medical disease
* Active infectious disease
* Previous pelvic radiation therapy
* Previous chemotherapy (prospective cohort)
* Patients with disease which can cause neutropenia
* Patients who will receive other targeted therapy or immunotherapy during adjuvant therapy (prospective cohort).
* Pregnant or lactating woman

Ages: 20 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Training cohort (prospective cohort): Patients with epithelial ovarian cancer who underwent staging operation or debulking surgery at university hospital and who are planned to receive adjuvant chemotherapy with paclitaxel and carboplatin.
  Validation cohort (retrospective cohort): Patients with epithelial ovarian cancer who received adjuvant chemotherapy with paclitaxel and carboplatin after staging operation or debulking operation.
Sampling Method: Probability Sample
Enrollment: 750 (Estimated)
Dates: Start 2012-09; Primary Completion 2018-05 (Estimated); Study Completion 2018-05 (Estimated)

PRIMARY OUTCOMES:
Risk prediction model for grade 3-4 chemotherapy induced neutropenia | 1 year

SECONDARY OUTCOMES:
The association between mannose-binding lectin 2 gene SNP and neutropenia | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Jeong-Yeol Park, M.D., Ph.D., Principal Investigator — Asan Medical Center
Locations (1):
- Department of Obstetrics and Gynecology, University of Ulsan College of Medicine, Asan Medical Center, Seoul, South Korea